CLINICAL TRIAL: NCT01822821
Title: Intravenous Acetaminophen Analgesia After Cardiac Surgery: A Randomized, Blinded, Controlled Superiority Trial
Brief Title: Pain Control After Cardiac Surgery Using Intravenous Acetaminophen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 13-269
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Pain
Keywords: Males or females; 18 years of age or older.; Non-emergency; cardiac surgery; midline sternotomy.
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Acetaminophen (Experimental): Patients will receive up to four doses of IV Acetaminophen (1000mg)every six hours after surgery along with standard PCA (patient controlled) opioids.
  Interventions: Drug: IV Acetaminophen
- Placebo (Placebo Comparator): Patients will receive up to four doses of IV placebo every six hours after surgery along with standard PCA (patient controlled) opioids.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Acetaminophen — Patients will receive up to four doses of IV Acetaminophen (1000mg)every six hours after surgery along with standard PCA (patient controlled) opioids.
  Other Names: 1000mg IV Acetaminophen
  Arms: IV Acetaminophen
Drug: Placebo — Patients will receive up to four doses placebo every six hours after surgery along with standard PCA (patient controlled) opioids.
  Other Names: inactive substance
  Arms: Placebo

SUMMARY:
Evaluate the efficacy of IV acetaminophen; compared to a placebo, in reducing opioid consumption and/or pain intensity scores after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* - Males or females 18 years of age or older.
* Non-emergency cardiac surgery via a midline sternotomy at Cleveland Clinic Main Campus.

Exclusion Criteria:

1. Redo cardiac surgery.
2. Combined CABG (Coronary Artery Bypass Graft)& valve replacement, multiple valve replacements, Ascending aortic or aortic arch surgery.
3. Weight < 50 Kg or Body mass index > 38 kg/m2.
4. Left ventricle EF ¡Ü 35% ,Right ventricular moderate or severe dysfunction.
5. Severe (3-4 +) Tricuspid Regurgitation.
6. Recent stroke (within 6 months).
7. Severe lung disease requiring home O2 therapy.
8. Preoperative renal insufficiency (Creatinine > 2.0) or on dialysis.
9. History of liver cirrhosis or active liver disease.
10. Chronic pain conditions controlled by preoperative opioid administration.
11. Known allergy to acetaminophen or fentanyl.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Negmeldeen Mamoun, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Acetaminophen | Placebo
Started | 75 | 75
Completed | 73 | 74
Not Completed | 2 | 1
Not completed — Eligible surgery cancelled | 1 | 1
Not completed — Other reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Placebo | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (14) | 59 (14) | 60.5 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Opioid Consumption
Description: Evaluate the noninferiority and efficacy of IV acetaminophen; compared to a placebo, in reducing opioid consumption a after cardiac surgery. Total opioid consumption is defined as the total amount amount of opioids administered to patients converted to mg morphine equivalents.
Time Frame: End of surgery through 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
mg morphine equivalents | 97 [58 to 136] | 117 [66 to 174]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Non-Inferiority or Equivalence — Noninferiority was tested using a noninferiority margin of 1.15; p = 0.08, Regression, Linear; ratio of geometric means = 0.89, 90% CI 1-sided [upper limit 1.06] — Ratio of geometric means (CI) for IV acetaminophen versus placebo was estimated as the exponentiated treatment effect parameter from a multivariable linear regression model on log opioid consumption adjusting for age and diabetes
Statistical Analysis 2: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.28, Regression, Linear; ratio of geometric means = 0.89, 95% CI 1-sided [upper limit 1.10] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Pain Intensity
Description: Evaluate the noninferiority and efficacy of IV acetaminophen; compared to a placebo, in reducing pain intensity scores after cardiac surgery. Pain scores were measured on the Numeric Rating scale, ranging from 0 to 10 (where 0 indicates no pain and 10 indicates the worst pain imaginable).
Time Frame: End of surgery through 24 hours after surgery
Population: All patients had at least one postoperative pain scores. Some patients did not have a pain score at particular time points if they were unavailable (e.g., at a test), unable to speak (e.g., intubated), asleep, or similar reasons. We report any available pain scores at each time they were collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
units on a scale
  overall pain scores | 3.1 (1.6) | 4.0 (1.4)
  4 hours after surgery: number analyzed (Participants) | 59 | 62
  4 hours after surgery | 4.6 (2.9) | 5.0 (3.1)
  6 hours after surgery: number analyzed (Participants) | 63 | 66
  6 hours after surgery | 3.5 (2.4) | 4.4 (2.4)
  8 hours after surgery: number analyzed (Participants) | 64 | 71
  8 hours after surgery | 3.2 (2.6) | 4.4 (2.3)
  12 hours after surgery: number analyzed (Participants) | 71 | 72
  12 hours after surgery | 2.4 (2.5) | 3.5 (2.6)
  16 hours after surgery: number analyzed (Participants) | 72 | 72
  16 hours after surgery | 3.0 (2.4) | 3.6 (2.4)
  20 hours after surgery: number analyzed (Participants) | 72 | 69
  20 hours after surgery | 2.9 (2.1) | 4.2 (2.0)
  24 hours after surgery: number analyzed (Participants) | 72 | 74
  24 hours after surgery | 2.5 (2.1) | 3.5 (2.0)
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Non-Inferiority or Equivalence — We assessed whether IV acetaminophen is noninferior to placebo using a noninferiority margin of 1.0; p < 0.001, Regression, Linear; Median Difference (Final Values) = -0.9, 90% CI 1-sided [upper limit -0.5] — Difference in overall postoperative pain score means based on a repeated measures linear regression model with an autoregressive correlation structure, adjusting for age, time, and diabetes
Statistical Analysis 2: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Linear; Mean Difference (Final Values) = -0.9, 95% CI 1-sided [upper limit -0.42] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Postoperative Nausea and Vomiting
Description: Incidence of any postoperative nausea and vomiting within 24 hours after surgery was collected.
Time Frame: End of surgery through 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
Participants | 16 | 21
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.35, Regression, Logistic; Risk Ratio (RR) = 0.76, 99.4% CI 2-sided [0.34 to 1.7] — Relative risk of PONV in IV acetaminophen versus placebo patients estimated from a multivariable logistic regression model using the log link and adjusting for age and diabetes

4. Secondary Outcome: Postoperative Sedation
Description: Postoperative sedation was assessed using the Richmond Agitation Sedation Scale (RASS). It ranges from -5 to +4, where -5 indicates no response to voice or physical stimulation and +4 indicates overtly combative or violent and immediate danger to staff. Lower the value, better the sedation.
Time Frame: Measured at 8, 16, and 24 hours after surgery
Population: RASS scores were not collected at certain time points if patients were not available (e.g., patient was away at a test) or if staff were not available.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
units on a scale
  8 hours after surgery: number analyzed (Participants) | 48 | 41
  8 hours after surgery | 0 [-1 to 0] | 0 [-1 to 0]
  16 hours after surgery: number analyzed (Participants) | 39 | 43
  16 hours after surgery | 0 [-1 to 0] | 0 [0 to 0]
  24 hours after surgery | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Analysis at 8 hours after surgery; Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 99.8% CI 2-sided [0 to 0] — Difference in medians of IV acetaminophen versus placebo patients based on Wilcoxon rank sum test and Hodges-Lehmann estimation of location shift
Statistical Analysis 2: Comparison: IV Acetaminophen vs Placebo; Analysis at 16 hours after surgery; Test type: Superiority or Other; p = 0.44, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 99.8% CI 2-sided [0 to 0] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: IV Acetaminophen vs Placebo; Analysis at 24 hours after surgery; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0, 99.8% CI 2-sided [0 to 0] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Duration of Mechanical Ventilation (Minutes)
Description: Evaluate whether IV acetaminophen reduced duration of Mechanical Ventilation.
Time Frame: End of surgery until the initial end of ventilation or date of death from any cause, whichever came first, assessed up to 1 week.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
minutes | 214 [143 to 345] | 190 [139 to 381]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.46, Regression, Linear; ratio of geometric means = 1.3, 99.4% CI 2-sided [0.52 to 3.20] — Outcome log-transformed to meet model assumptions. The treatment effect on duration of mechanical ventilation was assessed by use of the ratio of geometric means from a multivariable logistic regression models adjusting for age and diabetes

6. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Description: Evaluate whether IV acetaminophen reduced intensive care unit (ICU) Length of Stay.
Time Frame: End of surgery through discharge from ICU
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
hours | 214 [143 to 345] | 190 [139 to 381]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.38, Regression, Linear; ratio of geometric means = 0.93, 99.4% CI 2-sided [0.74 to 1.20] — Outcome log-transformed to meet model assumptions. The treatment effect on duration of ICU stay was assessed by use of the ratio of geometric means from a multivariable logistic regression models adjusting for age and diabetes

7. Secondary Outcome: Hospital Length of Stay
Description: Evaluate whether IV acetaminophen hospital length of stay
Time Frame: end of surgery through hospital discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
days | 6.2 [5.3 to 7.3] | 6.1 [5.1 to 7.2]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.12, Regression, Linear; ratio of geometric means = 1.1, 99.4% CI 2-sided [0.94 to 1.20] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Alanine Aminotransferase (ALT); U/L
Time Frame: Two days after surgery or date of death from any cause, whichever came first
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
U/L
  Overall ALT | 18 [15 to 23] | 19 [15 to 24]
  postoperative day 1 ALT | 18 [16 to 24] | 19 [15 to 25]
  postoperative day 2 ALT | 17 [14 to 22] | 18 [15 to 23]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.31, Regression, Linear; ratio of geometric means = 1.1, 99.4% CI 2-sided [0.9 to 1.2] — Outcome log-transformed to meet model assumptions. The treatment effect on ALT was assessed by use of the ratio of geometric means from a repeated measures multivariable logistic regression models adjusting for age and diabetes

9. Secondary Outcome: Aspartate Aminotransferase (AST); U/L
Time Frame: Two days after surgery or date of death from any cause, whichever came first
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
U/L
  Overall AST | 35 [30 to 45] | 33 [29 to 51]
  postoperative day 1 AST | 40 [32 to 54] | 40 [32 to 57]
  postoperative day 2 AST | 31 [24 to 42] | 31 [23 to 45]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.98, Regression, Linear; ratio of geometric means = 1.0, 99.4% CI 2-sided [0.8 to 1.2] — Outcome log-transformed to meet model assumptions. The treatment effect on AST was assessed by use of the ratio of geometric means from a repeated measures multivariable logistic regression models adjusting for age and diabetes

10. Secondary Outcome: Total Bilirubin (mg/dL)
Time Frame: Measured at 1 day and 2 days after surgery
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 73 | 74
mg/dL
  overall bilirubin | 0.7 [0.5 to 0.9] | 0.7 [0.5 to 0.8]
  postoperative day 1 bilirubin | 0.7 [0.5 to 1.0] | 0.7 [0.5 to 0.8]
  postoperative day 2 bilirubin | 0.6 [0.4 to 0.8] | 0.6 [0.4 to 0.8]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.40, Regression, Linear; ratio of geometric means = 1.1, 99.4% CI 2-sided [0.87 to 1.3] — Outcome log-transformed to meet model assumptions. The treatment effect on bilirubin was assessed by use of the ratio of geometric means from a repeated measures multivariable logistic regression models adjusting for age and diabetes

ADVERSE EVENTS:
Arm/Group | IV Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/74
Other Adverse Events (participants affected / at risk) | 0/73 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes